CLINICAL TRIAL: NCT06132243
Title: A Single-dose, Randomized, Open-label, Repeated Cross-over Pharmacokinetic Comparison Study of Two Formulations of Jaktinib Hydrochloride Tablets in Healthy Adult Volunteers Under Fasted Conditions
Brief Title: Comparative Study on Pharmacokinetics of Two Formulations of Jaktinib in Healthy Adults Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK037
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Subjects in the first sequence of the first cycle were administered with a test formulation (T) of 50 mg of Jaktinib on an empty stomach, while subjects in the second sequence were administered with a reference formulation (R) of 50 mg of Jaktinib on an empty stomach. The reference formulation (R) or test formulation (T) was administered alternately in the next periods.
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Reference Group (Active Comparator): Subjects in the first sequence of the first cycle were administered with a test formulation (T) of 50 mg of Jaktinib on an empty stomach, while subjects in the second sequence were administered with a reference formulation (R) of 50 mg of Jaktinib on an empty stomach. The reference formulation (R) or test formulation (T) was administered alternately in the next periods.
  Interventions: Drug: Jaktinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Orally, one tablet at a time
  Other Names: Jaktinib

SUMMARY:
To evaluate the pharmacokinetic Characteristics of two formulations of Jaktinib Hydrochloride Tablets in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age ≤ 45, male or female;
* Body weight: ≥50 kg for male, ≥45 kg for female; body mass index (BMI): 19.0-26.0 kg/m^2 (inclusive);
* Informed consent will be signed before the trial, and the content, process and possible adverse reactions of the trial will be fully understood;
* The volunteers should be able to communicate well with the researchers and understand and comply with the requirements of the study.

Exclusion Criteria:

* Participants who were enrolled in a clinical trial or used a study drug within 3 months before administration of the study drug;
* Participants with chronic or active gastrointestinal diseases such as esophageal disease, gastritis, gastric ulcer, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery within the past three years and still clinically relevant according to the investigator;
* Participants with definite diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, metabolic system and other diseases that require medical intervention or are not suitable for clinical trial (such as psychiatric history);
* With positive alcohol breath test;
* Volunteers may not be able to complete the study for other reasons or have other reasons for not participating in the study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) Of Jaktinib and its main metabolite ZG0244 | up to 48 hours
  Maximum Plasma Concentration (Cmax)
Jaktinib and its main metabolite ZG0244 AUC(0-t) | up to 48 hours
  Area under the concentration time curve from time 0 to time of the last quantifiable
Jaktinib and its main metabolite ZG0244 AUC(0-inf) | up to 48 hours
  Area under the concentration time curve from time 0 to infinity

SECONDARY OUTCOMES:
Jaktinib and its main metabolite ZG0244 Tmax | up to 48 hours
  Maximum Plasma Concentration (Tmax)
Jaktinib and its main metabolite ZG0244 t1/2 | up to 48 hours
  Half Life (t1/2)
Adverse events | Day 1 to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No